CLINICAL TRIAL: NCT03101696
Title: Determination of Coronarphysiological Parameters With the Method of Thermodillution
Status: Completed | Type: Observational
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Principal Investigator, Klinik für Kardiologie, Pneumologie und Angiologie, Dr. med. Florian Bönner, Heinrich-Heine University, Duesseldorf
Other Study IDs: 16-024
Record Dates: First submitted 2017-03-30; First posted 2017-04-05 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Stenosis of Unclear Hemodynamic Relevance
Keywords: coronary angiography; coronary conductance; hyperemia; regadenoson; fractional flow reserve; coronary flow reserve; index of microcirculatory resistance
MeSH Terms: conditions — Hyperemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The gold standard to induce coronary hyperemia for measurement of fractional flow reserve (FFR), coronary flow reserve (CFR) and index of microcirculatory resistance (IMR) is adenosine, but it exerts several side effects due to its unspecific action on adenosine receptors. The specific A2a-receptor agonist, regadenoson, has been shown to dilate coronary arteries and enables FFR measurements. The aim of the study was to evaluate whether simultaneous measurement of FFR, CFR and IMR is feasible, safe and effective within regadenoson-induced hyperemia.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR), coronary flow reserve (CFR) and the index of microcirculatory resistance (IMR) provide significant information on the conductance of coronary macro- and microcirculation.

FFR-based functional assessment of coronary artery disease has proven to be superior to purely morphologic assessment and thereby guides therapy decision. IMR is a pressure-temperature derived parameter for quantifying microcirculatory resistance, which has been proven to be relatively independent of epicardial stenosis severity when taking collateral flow into account. IMR is increased in patients with acute myocardial infarction and microvascular obstruction (MVO) as assessed by contrast-enhanced CMR and predicts left ventricular function and enddiastolic volumes at 6 month independently of initial infarct size.

Most interestingly, even in the absence of obstructive coronary artery disease, IMR is elevated in more than 20% of patients presenting with chest pain. The clinical meaning for this finding has to be elucidated.

FFR, CFR and IMR can only be measured under conditions of minimal coronary resistance with the need for coronary hyperemia. The current "gold standard" to induce hyperemia in the assessment of coronary conductance is adenosine. However, adenosine is known to cause side effects (bronchospasm and disturbances in atrioventricular conduction) due to its unselective action on all adenosine receptors. Besides that, adenosine requires a body weight adapted dosing and continuous infusion. However, alternative routes like intracoronary injection show good correlation compared with the intravenous route and side effects can be reduced. In contrast, regadenoson, a specific A2A receptor agonist, exhibits negligible side effects. It can be administered intravenously as a non-body weight adapted bolus via peripheral vein without the need for transfemoral delivery. Thus, patients with a transradial access for cardiac catheterization might benefit the most from inducing hypermedia via peripheral vein. It has already been shown that regadenoson increases coronary blood flow yielding comparable values for FFR and indexes of perfusion in SPECT. However, the duration and stability of regadenoson-induced hyperemia might be insufficient for a simultaneous measurement of FFR, CFR and IMR, which has not been tested so far.

The aim of the present study is to evaluate whether simultaneous measurement of the parameters FFR, CFR and IMR under regadenoson-induced hyperemia is feasible, safe and effective in patients with stable coronary artery disease undergoing a transradial procedure

ELIGIBILITY:
Inclusion Criteria:

Coronary angiography with indication of FFR measurement

* angiography without pathological results explaining the patients' symptoms
* intermediate stenosis (50-70%)

Exclusion Criteria:

* <18 years
* Hypersensitivity towards regadenoson
* hemodynamic instability
* severe hypotension
* acute myocardial ischemia
* AV block II-III

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with indication for FFR measurement due to a coronary artery stenosis of unclear hemodynamic relevance
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-02-05 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
fractional flow reserve (FFR) | Baseline
  Description: the proximal aortic (Pa) and distal arterial pressure (Pd) are recorded and RadiAnalyzer Xpress™ control unit automatically calculates FFR as Pd/Pa

SECONDARY OUTCOMES:
coronary flow reserve | Baseline
  The RadiAnalyzer Xpress™ calculates CFR as Tmnr/Tmnh
index of microcirculatory resistance | Baseline
  Using the derived Pd and transit mean times under hyperemia (Tmnh), it will be calculated apparent IMR as Pd×Tmnh. All IMR values are also corrected by Yong's formula (IMRcorr=Pa×Tmnh×([1.35×Pd/Pa]-0.32) to adjust for the influence of collateral flow.

CONTACTS AND LOCATIONS:
Overall Officials: Malte Kelm, MD, Study Chair — Division of Cardiology, Pulmonary Disease and Vascular Medicine
Locations (1):
- Division of Cardiology, Pulmonary Disease and Vascular Medicine, Düsseldorf, Germany

IPD SHARING:
Plan to Share IPD: Yes